CLINICAL TRIAL: NCT04905485
Title: Developing a Model to Better Predict Diabetes and/or Risk of Developing Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: V136 (VIOME-001 v5.0)
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Type 2; Diabetes; Pre-diabetes
Keywords: Viome; Diabetes Type 2; Diabetes; Pre-diabetes; VPNP; Nutrition; Supplements; Precision
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Participants all received diet and supplement recommendations based on their microbiome results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): All participants received the intervention in this trial. They received recommendations on their diets and supplements based on their results of microbiome expression.
  Interventions: Behavioral: VIOME Precision Nutrition Program

INTERVENTIONS:
Behavioral: VIOME Precision Nutrition Program — Precision diet and supplement recommendations based on participants' microbiome results.
  Other Names: VPNP

SUMMARY:
Participants who were previously Viome costumers who signed informed consent to participate and self reported type 2 diabetes or pre-diabetes were enrolled. They provided stool samples to VIOME and were provided with precision diet and supplement recommendations. The information obtained from this study is used to train a model to predict diabetes and/or risks of developing diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Viome customer
* GI test collected at home using Viome test kit
* US citizen
* 18+ years old
* Is not participating in any other Viome study
* Must have answered the following on-boarding question with the indicated answer:

"Do you or did you ever have diabetes or prediabetes?"

* Signed and dated informed consent prior to any trial-specific procedures are performed
* Able to speak and read English
* Willing and able to follow the trial instructions

Exclusion Criteria:

* Unable/unwilling to complete the informed consent form and the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2912 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in VIOME's Type 2 diabetes risk score | ~3 months
  "Type 2 diabetes risk score" is computed using Viome's molecular data from stool and HBA1C level self reported. The risk score is 1-100. 1 Indicates a low chance of developing T2D and 100 indicates a high chance of developing T2D.

CONTACTS AND LOCATIONS:
Overall Officials: Guruduth Banavar, PhD, Principal Investigator — Viome
Locations (1):
- Viome Research Institute, Bothell, Washington, United States

IPD SHARING:
Plan to Share IPD: No